## OFFICIAL TITLE OF THE STUDY: LVA2017

NCT ID not yet assigned

DATE OF THE DOCUMENT: January 26th 2018

## Statistical analysis

The correlation between the time from onset of lymphedema and primary and secondary outcomes will be investigated with Cox proportional hazard model

Differences in outcome measures between recent (<1 year) and long standing lymphedema will be investigated using Generalized Linear Models using gaussian family and identity link.

When more than one sample from the same patient is present, the patient will be included in the model as a random effect variable.

A p value of 0.05 or less for a two tails distribution will be considered statistically significant.

Data is presented as M  $\pm$  robust SE

All the analyses will be performed using Stata vers. 12 (Stata Corp, College Station, TX)